CLINICAL TRIAL: NCT03261726
Title: Maintaining Cochlear Patency After VIIIth Nerve Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No subjects were enrolled.
Sponsor: Henry Ford Health System (Other)
Collaborators: Med-El Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB# 1040241
Record Dates: First submitted 2017-08-20; First posted 2017-08-25 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2021-03

CONDITIONS: Acoustic Neuroma; Labyrinthitis Ossificans; Profound Hearing Impairment
Keywords: unilateral deafness; acoustic neuroma; cochlear implant
MeSH Terms: conditions — Neuroma, Acoustic; Hearing Loss, Unilateral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- MedEl Test Electrode Placer (Experimental): MedEl Test Electrode Placed at VIIIth nerve tumor resection
  Interventions: Device: MedEl Test Electrode Placer

INTERVENTIONS:
Device: MedEl Test Electrode Placer — This study uses a sterile dummy (i.e., not working) cochlear implant electrode inserted at the time of tumor removal to keep the inner ear from scarring or filling with bone. The significance of this to you is that if you ever become eligible for a cochlear implant sometime after surgery, it may be possible to remove the dummy and insert a functioning cochlear implant.

SUMMARY:
Tumors arising from the VIIIth Nerve (vestibulo-cochlear nerve) typically present with progressive unilateral hearing loss and tinnitus. VIIIth Nerve tumors with documented growth on serial MRI scans typically lead to deafness in the affected ear over time. Radiation (Gamma Knife® or stereotactic radiosurgery) may preserve hearing in ~80% while surgery (middle cranial fossa or retrosigmoid approach) may preserve hearing in 16 - 40% of small tumors, although initial hearing preservation by both modalities may fail over time. Surgical resection via the translabyrinthine approach is the safest way to remove many of these tumors, but involves loss of all hearing. In all treatment modalities, the vascular supply (the labyrinthine artery, a terminal branch of AICA with no collaterals) to the cochlea is at risk. After devascularization, the cochlea frequently fills with fibrous tissue or ossifies (labyrinthitis ossificans), making it impossible to place a cochlear implant should it be required later. The incidence of this is 46% in our patients. This study seeks to determine the feasibility of preserving the cochlear duct with an obdurator so that patients undergoing translabyrinthine removal of VIIIth nerve tumors may retain the option of a cochlear implant at a later time.

ELIGIBILITY:
Inclusion Criteria:

* patients of all ages with unilateral or bilateral acoustic neuromas who face loss of hearing in 1 ear from surgical removal via a translabyrinthine approach.
* patients do not meet criteria for conventional cochlear implantation or auditory brainstem implantation.
* tumor removal must allow preservation of the auditory division of the VIIIth cranial nerve.
* the patient must be willing to undergo preoperative S pneumococcus immunization protocol recommended by the US CDC immunization recommendations for cochlear implant patients.

Exclusion Criteria:

* inability to preserve the auditory division of the VIIIth cranial nerve during tumor removal ossification or fibrosis of the cochlea found on preoperative imaging (CT or MRI) that precludes cochlear implantation.
* active middle ear disease.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-04 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-03-04 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events related to implanted insertion electrode | One year postoperatively
  Office visits and MRI monitoring:
  1. 2 - 3 weeks after surgery: Routine post-operative visit for wound care. I. Document integrity and appearance of the eardrum. II. Document wound integrity and appearance.
  2. 3 - 4 months after surgery: Monitoring MRI with and without contrast of the inner ear/internal auditory canals with routine post-operative visit. I. Document integrity and appearance of the eardrum. II. Document wound integrity and appearance. III. Document appearance of the cochlea on heavily T2-weighted images.
  3. Study Endpoint: 1 year after surgery. Repeat MRI with and without contrast of the inner ear/internal auditory canals. I. Document integrity and appearance of the eardrum. II. Document wound integrity and appearance. III. Document appearance of the cochlea on heavily T2-weighted images.

SECONDARY OUTCOMES:
Presence or absence of fluid in the cochlea | 3- 4 months and 1 year after tumor removal and implantation of the insertion electrode
  Appearance of the implanted cochlea on heavily T2-weighted monitoring MRI 3-4 months after surgery and 1 year after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Eric W Sargent, MD, Principal Investigator — Ascension Providence Hospital
Locations (1):
- The Michigan Ear Institute, Farmington Hills, Michigan, United States

IPD SHARING:
Plan to Share IPD: No